CLINICAL TRIAL: NCT00317330
Title: A Randomized Trial of DOTS Versus Enhanced DOTS for Community Control of Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-581; ICIDR#1
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2006-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; Pyrazinamide; Rifampin

INTERVENTIONS:
Drug: Isoniazid
Drug: Pyrazinamide
Drug: Rifampin

SUMMARY:
This study will test the effectiveness of two different tuberculosis (TB) prevention strategies, DOTS or DOTS-A. DOTS is the current prevention strategy for TB. DOTS-A is an enhanced prevention strategy that will screen household members of individuals diagnosed with active TB and will provide enhanced treatment as needed. The study will be conducted in 8 communities located in Rio de Janeiro. Study participants will include 6400 males and females of all ages, including active TB patients and their household contacts. Patients with TB identified for treatment at the Health Clinics of 8 urban communities will be eligible. The communities will be assigned to 1 of the 2 prevention strategies, DOTS or DOTS-A. After 4 years, the information gathered during the study will be used to determine the incidence of TB in these communities to see which prevention strategy was more effective in decreasing TB.

DETAILED DESCRIPTION:
This will be a single site, prospective, community-randomized trial to study the effectiveness for two TB prevention strategies on the community incidence of TB: DOTS versus Enhanced DOTS (DOTS-Ampliado, or DOTS-A). DOTS-A will add intensive screening of household contacts of active TB cases and the provision of TB treatment or prophylaxis as needed to the standard DOTS regimen. Adult contacts in the DOTS-A communities will be offered enrollment into a randomized clinical trial comparing rifapentine/isoniazid preventive therapy to rifampin/pyrazinamide. Subjects will be recruited from TB cases identified for treatment at the Health Clinics of eight urban communities. These communities will be matched and randomly assigned to receive either DOTS or DOTS-A strategy. The change in the incidence of TB in the two groups of communities will be measured after a 4-year period to determine whether DOTS-A strategy significantly reduces the incidence of TB compared to DOTS alone.

ELIGIBILITY:
Inclusion Criteria:

Cases will include:

1. Any age male or female with new or recurrent diagnosis of TB
2. Willingness and ability to adhere to study medications and protocol procedures.
3. Willingness to provide signed informed consent or signed informed consent/assent provided by parent or legal guardian.

Contacts will include:

1. Male or female living in household of a pulmonary TB case, at high risk for developing TB (but without evidence for active TB).
2. High-risk household contacts will be defined as those who are:

   * HIV seropositive, regardless of the results of initial tuberculin skin test (TST)
   * TST positive at the time of the first household evaluation. TST positivity will be defined as greater than or equal to 5 mm induration of 5 TU of PPD using the Mantoux method, read between 48 and 72 hours after application.
   * TST negative at the time for the first household evaluation and TST positive at the time of the second household evaluation 3 months later.
   * Willingness to provide signed informed consent or signed informed consent/assent provided by parent or legal guardian.

Exclusion Criteria:

Contacts will be excluded from preventive therapy if:

1. Current active clinical tuberculosis-confirmed or suspected
2. History of sensitivity/intolerance to any of the study medications
3. Evidence of acute hepatitis
4. History or laboratory evidence of cirrhosis
5. Pregnant females (treatment of latent infection will be deferred)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6400
Dates: Start 2004-12; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Locations (1):
- Municipal Health Department, Rio de Janeiro, Brazil